CLINICAL TRIAL: NCT04932785
Title: To Assess the Comparative Efficacy of Full Calorie Regular Diet (RD) Versus Clear Liquid Diet (CLD) on Length of Hospital Stay (LOHS) for Mild to Moderate Acute Pancreatitis (AP)
Brief Title: Regular vs. Clear Liquid Diet for Mild to Moderate Acute Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, James Buxbaum, Chief of Gastroenterology Los Angeles County + University of Southern California, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-20-00375
Record Dates: First submitted 2021-06-07; First posted 2021-06-21 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Pancreatitis; Diet, Food, and Nutrition; Diet; Pancreatic Disease; Enteral Nutrition
MeSH Terms: conditions — Pancreatitis; Pancreatic Diseases | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular Diet (Active Comparator): Patient randomized to regular diet will begin with a regular diet.
  Interventions: Other: Regular diet
- Clear Liquid Diet (Active Comparator): Patient randomized to clear liquid diet will begin with a clear liquid diet.
  Interventions: Other: Clear Liquid Diet

INTERVENTIONS:
Other: Regular diet — Regular diet
  Arms: Regular Diet
Other: Clear Liquid Diet — Clear Liquid Diet
  Arms: Clear Liquid Diet

SUMMARY:
Acute pancreatitis is among the most common gastroenterology diagnosis in the United States, and represents a large economic burden to the United States health system. While recent guidelines agree early feeding shortens length of stay, these guidelines fail to provide recommendations on optimal diet to start leaving diet type to clinician discretion. Therefore, the aim is to assess the comparative efficacy of full calorie regular diet (RD) versus clear liquid diet (CLD) on length of hospital stay (LOHS) for mild to moderate acute pancreatitis (AP). The study population will target mild to moderate acute pancreatitis patients who can tolerate eating in a single institution. The primary end point will focus on LOHS, and secondary end points will include Pancreatic Activity Scoring System, side effects and readmission.

DETAILED DESCRIPTION:
Purpose: To assess the comparative efficacy of initial full calorie regular diet (RD) versus clear liquid diet (CLD) on length of hospital stay (LOHS) for mild to moderate acute pancreatitis (AP).

Study Design:

Patients presenting to the Los Angeles County Hospital with mild to moderate acute pancreatitis are eligible and are the focus population of this study. Diagnosis and severity classification will be according to the Revised Atlanta classification and Modified Marshal Score. Patients will require fulfillment of 2 of 3 criteria: amylase or lipase greater than 3 times the upper limit of normal, classic epigastric abdominal pain, or unequivocal imaging consistent with acute pancreatitis.

Patients within the inclusion and exclusion parameters will be randomized to RD vs. CLD within 16 hours of diagnosis of pancreatitis. Randomization will be performed using a random sequence algorithm with concealed allocation. The provision of diet in the emergency department prior to randomization will be recorded but not impact randomization strategy.

Following randomization, the diet of RD vs. CLD will begin as soon as patient expresses an appetite and willingness to eat. The patients will be assessed within 24 hours for hunger and interest in initiating oral feeding which accords with the 2018 recommendations of the American Gastroenterology Association for the management of acute pancreatitis.

The diet algorithm will be randomization to a 1:1 of full regular diet versus clear liquid diet per the Los Angeles County + University of Southern California nutrition department. This nutritional composition is confirmed by the in-house dietician and nutrition department. Regular diet will reflect the U.S. Department of Health and Human Services Dietary guidelines for 2015-202013 and meets recommendations of the International Consensus Guidelines for Nutrition Therapy for Pancreatitis. Fat content is modest in both groups; it is set at 20-35% of caloric intake for regular diet and 15-20% for clear liquid diet. Patients with diabetes mellitus will received modified versions of the regular or clear diet to reflect American Diabetes Association (ADA) requirements. This will be the standard of care composition provided to all patients at Los Angeles County + University of Southern California Medical Center with diabetes deemed by their providers to have a diet modified for diabetes (ADA) diet.

A complete history and physical exam will be taken at time of admission within 24 hours during time of enrollment. Then at 48 hours, 72 hours, and every day until discharge, the patient will have a targeted history including oral tolerance, pain and pain medication requirement, and baseline and changes in Pancreatic Activity Scoring System (PASS). The percent of completed diet per meal will also be recorded. At one week, patients will be contacted for symptom relapse check up by phone and at thirty days, the electronic record will be reviewed to capture possible readmissions. While patients and the study team will be unblinded following discharge, a blinded coordinator will use the length of stay function to capture the primary endpoint which is length of hospitalization.

Pain and pain medications are automatically documented in the Electronic Medical Record(EMR) for monitoring and quantification. A Wong-Baker Pain (FACES) scale is the current validated pain score used by nursing staff. Pain is recorded on a pain scale from 0-10 that matches prior landmark and contemporary studies of acute pancreatitis. Quantification of pain medication by both acetaminophen and morphine equivalents will be recorded in data collection sheets.

If patients have oral intolerance or ileus, their diet will be managed at the discretion of their treating physicians and recorded by the study team. It will be recommended that diets remain consistent and titrated in quantity per physician and patient preference; however, if there is a physician preference to change to a different diet type this will be recorded and the patient will be included in the intention to treat analysis

For severe pancreatitis that develops following enrollment, nutritional management (whether nasal jejunal tube or total parenteral nutrition) will be managed per the primary team and patients will similarly be included in the intention to treat analysis.

Gallstone pancreatitis will be diagnosed by findings of elevated or fluctuating liver enzyme tests and biliary imaging abnormalities including cholelithiasis or ductal dilation. For patients with gallstone pancreatitis who will undergo same admission cholecystectomy, patients will have diet prescribed per assigned randomization but will be made nothing by mouth (NPO) at the discretion of the surgical team in anticipation of the operation. Integration of surgery into the hospitalization may impact length of stay. Therefore, randomization will be stratified by presence of gallstone versus non-gallstone pancreatitis.

Additionally, the study protocol will not impact other strategies/treatments to manage pancreatitis. For example, alcohol counseling will be provided to those whose pancreatitis is related to heavy alcohol use regardless of randomization or the study.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Presentation with acute pancreatitis as defined by two of three criterion per the Revised Atlanta Criteria guidelines: (a) Amylase or lipase > 3x the upper limit of normal, b) Classical abdominal pain, c) Ultrasound or computed tomography of unequivocal pancreatitis. Such radiographic findings include swelling, edema, or heterogeneity of the gland or peripancreatic fluid or stranding

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Incarcerated patients
3. Patients < 18 years of age
4. Patient unable or unwilling to give informed consent
5. Patients transferred from another hospital
6. The possibility of poor oral intake for reasons other than acute pancreatitis (e.g. intubation, failure to pass an indicated swallow study for aspiration risk, anorexia secondary to active malignancy, etc)
7. Surgical intervention for infected pancreatic necrosis or pancreatic hemorrhage
8. Chronic pancreatitis based on radiographic evidence
9. Severe pancreatitis based on Revised Atlanta Criteria. Under Revised Atlanta Criteria, patients will be excluded if they have a composite Modified Marshall >2
10. Etiologies of hypertriglyceridemia, trauma and autoimmune pancreatitis will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-18 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Length of Hospitalization Stay | From date of randomization until the date of discharge, assessed up to 24 months
  Length of Hospitalization Stay will be measured as defined as from time of admission to time of discharge for regular diet vs. clear liquid diet

SECONDARY OUTCOMES:
Oral Intolerance | From date of randomization until the date of discharge, assessed up to 24 months
  Proportion who cannot tolerate assigned diet requiring cessation or change due to worsened nausea, vomiting and pain
Intensive Care Unit admission and interventions | From date of randomization until the date of discharge, assessed up to 24 months
  Intensive Care Unit admission and intervention including intubation and vasopressors
Local complications | From date of randomization until the date of discharge, assessed up to 24 months
  Local complications including pancreatic necrosis, abscess, or pseudocysts
Development of severe pancreatitis | From date of randomization until the date of discharge, assessed up to 24 months
  Development of severe pancreatitis as defined by the Revised Atlanta Classification (persistent single or multiple organ failure at >48 hours)
Development of severe pancreatitis | From date of randomization until the date of discharge, assessed up to 24 months
  Development of severe pancreatitis as defined by the Modified Marshall Score (Score 0-4, with 4 being most severe and worse outcome)
Change in Pancreatic Activity Scoring System Score | From date of randomization until the date of discharge at 24, 48, 72 hours and at discharge, assessed up to 24 months
  Change in Pancreatic Activity Scoring System Score, from 0 to >250 (max score, where a max score is worse)
Calorie and fat intake | From date of randomization until the date of discharge, assessed up to 24 months
  Calorie and fat intake per group based on percent finished meal documented by nursing staff at 24, 48, and 72 hours.
30 day hospital readmission | From date of discharge to 30 days after discharge
  Hospital readmission within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: James Buxbaum, MD, Principal Investigator — Principal Investigator
Locations (1):
- LAC+USC Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Background] Peery AF, Crockett SD, Murphy CC, Lund JL, Dellon ES, Williams JL, Jensen ET, Shaheen NJ, Barritt AS, Lieber SR, Kochar B, Barnes EL, Fan YC, Pate V, Galanko J, Baron TH, Sandler RS. Burden and Cost of Gastrointestinal, Liver, and Pancreatic Diseases in the United States: Update 2018. Gastroenterology. 2019 Jan;156(1):254-272.e11. doi: 10.1053/j.gastro.2018.08.063. Epub 2018 Oct 10. PMID 30315778
- [Background] Jenkins A, Shapiro J. Clinical Guideline Highlights for the Hospitalist: Initial Management of Acute Pancreatitis in the Hospitalized Adult. J Hosp Med. 2019 Dec 1;14(12):764-765. doi: 10.12788/jhm.3324. Epub 2019 Oct 23. PMID 31634105
- [Background] Yadav D, Lowenfels AB. The epidemiology of pancreatitis and pancreatic cancer. Gastroenterology. 2013 Jun;144(6):1252-61. doi: 10.1053/j.gastro.2013.01.068. PMID 23622135
- [Background] Larino-Noia J, Lindkvist B, Iglesias-Garcia J, Seijo-Rios S, Iglesias-Canle J, Dominguez-Munoz JE. Early and/or immediately full caloric diet versus standard refeeding in mild acute pancreatitis: a randomized open-label trial. Pancreatology. 2014 May-Jun;14(3):167-73. doi: 10.1016/j.pan.2014.02.008. Epub 2014 Mar 14. PMID 24854611
- [Background] Jacobson BC, Vander Vliet MB, Hughes MD, Maurer R, McManus K, Banks PA. A prospective, randomized trial of clear liquids versus low-fat solid diet as the initial meal in mild acute pancreatitis. Clin Gastroenterol Hepatol. 2007 Aug;5(8):946-51; quiz 886. doi: 10.1016/j.cgh.2007.04.012. Epub 2007 Jul 5. PMID 17613280
- [Background] Sathiaraj E, Murthy S, Mansard MJ, Rao GV, Mahukar S, Reddy DN. Clinical trial: oral feeding with a soft diet compared with clear liquid diet as initial meal in mild acute pancreatitis. Aliment Pharmacol Ther. 2008 Sep 15;28(6):777-81. doi: 10.1111/j.1365-2036.2008.03794.x. PMID 19145732
- [Background] Li J, Xue GJ, Liu YL, Javed MA, Zhao XL, Wan MH, Chen GY, Altaf K, Huang W, Tang WF. Early oral refeeding wisdom in patients with mild acute pancreatitis. Pancreas. 2013 Jan;42(1):88-91. doi: 10.1097/MPA.0b013e3182575fb5. PMID 22836861
- [Background] Eatock FC, Chong P, Menezes N, Murray L, McKay CJ, Carter CR, Imrie CW. A randomized study of early nasogastric versus nasojejunal feeding in severe acute pancreatitis. Am J Gastroenterol. 2005 Feb;100(2):432-9. doi: 10.1111/j.1572-0241.2005.40587.x. PMID 15667504
- [Background] Rajkumar N, Karthikeyan VS, Ali SM, Sistla SC, Kate V. Clear liquid diet vs soft diet as the initial meal in patients with mild acute pancreatitis: a randomized interventional trial. Nutr Clin Pract. 2013 Jun;28(3):365-70. doi: 10.1177/0884533612466112. Epub 2012 Dec 13. PMID 23239793
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Crockett S, Falck-Ytter Y, Wani S, Gardner TB. Acute Pancreatitis Guideline. Gastroenterology. 2018 Mar;154(4):1102. doi: 10.1053/j.gastro.2018.02.029. Epub 2018 Mar 2. No abstract available. PMID 29501369
- [Background] American Diabetes Association. 15. Diabetes Care in the Hospital: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S193-S202. doi: 10.2337/dc20-S015. PMID 31862758
- [Background] Moraes JM, Felga GE, Chebli LA, Franco MB, Gomes CA, Gaburri PD, Zanini A, Chebli JM. A full solid diet as the initial meal in mild acute pancreatitis is safe and result in a shorter length of hospitalization: results from a prospective, randomized, controlled, double-blind clinical trial. J Clin Gastroenterol. 2010 Aug;44(7):517-22. doi: 10.1097/MCG.0b013e3181c986b3. PMID 20054282
- [Background] Buxbaum J, Quezada M, Chong B, Gupta N, Yu CY, Lane C, Da B, Leung K, Shulman I, Pandol S, Wu B. The Pancreatitis Activity Scoring System predicts clinical outcomes in acute pancreatitis: findings from a prospective cohort study. Am J Gastroenterol. 2018 May;113(5):755-764. doi: 10.1038/s41395-018-0048-1. Epub 2018 Mar 15. PMID 29545634
- [Background] Horibe M, Iwasaki E, Nakagawa A, Matsuzaki J, Minami K, Machida Y, Tamagawa H, Takimoto Y, Ueda M, Katayama T, Kawasaki S, Matsushita M, Seino T, Fukuhara S, Kanai T. Efficacy and safety of immediate oral intake in patients with mild acute pancreatitis: A randomized controlled trial. Nutrition. 2020 Jun;74:110724. doi: 10.1016/j.nut.2020.110724. Epub 2020 Jan 15. PMID 32200266
- [Background] Khan S, Ranjha WA, Tariq H, Nawaz H. Efficacy of early oral refeeding in patients of mild acute pancreatitis. Pak J Med Sci. 2017 Jul-Aug;33(4):899-902. doi: 10.12669/pjms.334.12338. PMID 29067062
- [Background] Greenberg JA, Hsu J, Bawazeer M, Marshall J, Friedrich JO, Nathens A, Coburn N, May GR, Pearsall E, McLeod RS. Clinical practice guideline: management of acute pancreatitis. Can J Surg. 2016 Apr;59(2):128-40. doi: 10.1503/cjs.015015. PMID 27007094
- [Background] Yokoe M, Takada T, Mayumi T, Yoshida M, Isaji S, Wada K, Itoi T, Sata N, Gabata T, Igarashi H, Kataoka K, Hirota M, Kadoya M, Kitamura N, Kimura Y, Kiriyama S, Shirai K, Hattori T, Takeda K, Takeyama Y, Hirota M, Sekimoto M, Shikata S, Arata S, Hirata K. Japanese guidelines for the management of acute pancreatitis: Japanese Guidelines 2015. J Hepatobiliary Pancreat Sci. 2015 Jun;22(6):405-32. doi: 10.1002/jhbp.259. Epub 2015 May 13. PMID 25973947
- [Background] Working Party of the British Society of Gastroenterology; Association of Surgeons of Great Britain and Ireland; Pancreatic Society of Great Britain and Ireland; Association of Upper GI Surgeons of Great Britain and Ireland. UK guidelines for the management of acute pancreatitis. Gut. 2005 May;54 Suppl 3(Suppl 3):iii1-9. doi: 10.1136/gut.2004.057026. No abstract available. PMID 15831893
- [Background] Mirtallo JM, Forbes A, McClave SA, Jensen GL, Waitzberg DL, Davies AR; International Consensus Guideline Committee Pancreatitis Task Force. International consensus guidelines for nutrition therapy in pancreatitis. JPEN J Parenter Enteral Nutr. 2012 May;36(3):284-91. doi: 10.1177/0148607112440823. Epub 2012 Mar 28. PMID 22457421
- [Background] Working Group IAP/APA Acute Pancreatitis Guidelines. IAP/APA evidence-based guidelines for the management of acute pancreatitis. Pancreatology. 2013 Jul-Aug;13(4 Suppl 2):e1-15. doi: 10.1016/j.pan.2013.07.063. PMID 24054878
- [Background] Meier R, Beglinger C, Layer P, Gullo L, Keim V, Laugier R, Friess H, Schweitzer M, Macfie J; ESPEN Consensus Group. ESPEN guidelines on nutrition in acute pancreatitis. European Society of Parenteral and Enteral Nutrition. Clin Nutr. 2002 Apr;21(2):173-83. doi: 10.1054/clnu.2002.0543. No abstract available. PMID 12056792